CLINICAL TRIAL: NCT02240264
Title: Food2Learn: Effect of Omega-3 LCPUFA Intervention on Learning, Cognition, Behaviour and Visual Processing.
Brief Title: Effect of Omega-3 LCPUFA Intervention on Learning, Cognition, Behaviour and Visual Processing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Open University (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government); Aker BioMarine Human Ingredients AS (Industry); Omegametrix GmbH (Unknown); Metrisquare (Unknown)
Responsible Party: Principal Investigator, Dr. Renate de Groot, Chair Brain, Lifestyle, and Learning Program, Open University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Food2Learn; 13-T-115 (Other: METC Atrium-Orbis-Zuyd)
Record Dates: First submitted 2014-09-05; First posted 2014-09-15 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Cognitive Function; Academic Performance; Mental Health
Keywords: Omega-3 fatty acids; Cognitive function; Academic performance; Mental health; Eye tracking; Krill oil; LCPUFA
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Krill oil capsules (Active Comparator): Capsules containing krill oil rich in omega-3 fatty acid's.
  Dietary supplements (krill oil) are provided by Aker BioMarine Antarctic AS equalling almost the daily recommended amount of 450 mg of EPA/DHA intake per day.
  Addendum 25-4-2016: In the Original protocol a dose adjustment after 3 months according to Omega-3 Index was to be executed. As no participant achieved the target Omega-3 Index the dosage was adjusted to 800mg DHA + EPA per day for all participants. The also led to the decision to increase the starting dosage of cohort II to 800mg DHA+ EPA.
  Interventions: Dietary Supplement: Krill oil capsules
- Placebo (Placebo Comparator): Capsules containing a fatty acid mixture that reflects the fatty acid composition of the average European diet.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Krill oil capsules — 1 year supplementation with Krill oil provided by Aker BioMarine Antarctic AS equalling almost the daily recommended amount of 450 mg of EPA/DHA intake per day.
  Arms: Krill oil capsules
Dietary Supplement: Placebo — Capsules containing a fatty acid mixture that reflects the fatty acid composition of the average European diet.
  Arms: Placebo

SUMMARY:
The brain is primarily developed in the third trimester of pregnancy, but continues maturing through the late twenties, especially the prefrontal cortex. Omega-3 long-chain polyunsaturated fatty acids (LCPUFA) are important structural components of neural cell membranes, influence membrane fluidity and signal transduction, and thus learning, cognition and behaviour. Levels of omega-3 LCPUFA have been found to be low in individuals with limitations in these complex brain functions. Previous studies suggested that such functions could be improved by increasing LCPUFA. The adolescent brain, however, has been largely neglected. This study investigates the effect of one-year daily omega-3 LCPUFA supplementation, in particular krill oil, in healthy 14-15 year old adolescents in lower general secondary education (MAVO/VMBO) on learning, cognition, and behaviour. The majority of the omega-3 PUFA in krill oil is incorporated into phospholipids, favouring tissue uptake of its omega-3 PUFA. In a double blind, randomised controlled trial, 300 adolescents preselected from a population of 700 adolescents with low omega-3 index (<5%) will receive daily omega-3 LCPUFA supplementation or matching placebo. The omega-3 LCPUFA dose will be adjusted individually to reach a target level of 8-11%. The effects on learning (academic achievement, objective cognitive performance), behaviour (mood, self-esteem, motivation, goal-orientation, absenteeism), and in a subsample cognitive processes, in particular perceptual processes measured by eye-tracking will be evaluated after 6, 12, and 24 months. This study will yield important insights in the effects of omega-3 LCPUFA supplementation, a safe intervention, on a large variety of complex brain functions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents aged 14-15 years.
* In lower general secondary education (MAVO/VMBO).

Exclusion Criteria:

* Suffering from hemophilia (blood clotting disorder).
* Allergic to (shell)fish.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 266 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | 12 months
  Neuropsychological tests covering seceral executive functions (LDST, D2, CST, Stroop, Digit Span).

SECONDARY OUTCOMES:
Eye tracking | 12 months
  Two types of eye tracking parameters will be calculated, namely basic parameters and paragraph-related parameters. Basic parameters are number of blinks, number of fixations, total duration of fixations, average fixation duration, average dispersion of fixation positions, average saccadic amplitude, and average saccadic velocity. Moreover, we will calculate eye tracking measures per paragraph, namely time spent on each paragraph (number and duration of fixations), time elapsed until first looking at a paragraph, and amount of times going back to a paragraph (revisits).
Academic achievement | 12 months
  Grade point average for Dutch, English and mathematics and standardized mathematics test scores (AMN).
Behaviour: absenteeism, motivation (MSLQ), Mood (CES-D), Self-esteem | 12 months
  Absenteeism, motivation (MSLQ), Mood (CES-D), Self-esteem
Sleep duration and sleep quality | 12 months
  Sleep duration measured using ActivPAL and diary, Sleep quality determined using the adolescent sleep wake scale (ASWS) and the adolescent sleep hygiene scale (ASHS).

CONTACTS AND LOCATIONS:
Overall Officials: Renate de Groot, PhD, Principal Investigator — Open University
Locations (17):
- Netherlands (17):
  - Canisius College, Nijmegen, Gelderland
  - MAVO Roermond, Roermond, Limburg
  - De Nassau, Breda, North Brabant
  - Graaf Engelbrecht, Breda, North Brabant
  - Newman College, Breda, North Brabant
  - Dr.Knippenberg College, Helmond, North Brabant
  - Stabrecht College, Geldrop
  - Graaf Huyn College, Geleen
  - Scholengemeenschap Sophianum, Gulpen
  - Citaverde, Heerlen
  - Grotius College, Heerlen
  - Sintermeertencollege, Heerlen
  - Beroepscollege Holz, Kerkrade
  - Bouwens van der Boijecollege, Panningen
  - DaCapo College, Sittard
  - Stella Maris College, Valkenburg
  - Colllege Den Hulster, Venlo

REFERENCES:
- [Derived] van der Wurff IS, von Schacky C, Berge K, Kirschner PA, de Groot RH. A protocol for a randomised controlled trial investigating the effect of increasing Omega-3 index with krill oil supplementation on learning, cognition, behaviour and visual processing in typically developing adolescents. BMJ Open. 2016 Jul 8;6(7):e011790. doi: 10.1136/bmjopen-2016-011790. PMID 27401364